CLINICAL TRIAL: NCT05786482
Title: Evidence Based Mental Wellness Programming Online for Adults Across Chronic Physical Conditions (EMPOwer) Randomized Controlled Trial
Brief Title: Evidence Based Mental Wellness Programming Online for Adults Across Chronic Physical Conditions
Acronym: EMPOwer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00122568
Record Dates: First submitted 2023-03-09; First posted 2023-03-27 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Primary Biliary Cholangitis; Heart Failure; Digestive Diseases; Women Who Have Experienced a Cardiac Event; Cirrhosis, Liver; Post-Transplant; Cancer; Chronic Kidney Diseases; Other Chronic Physical Condition
Keywords: Mind Body Wellness; Depression; Anxiety; Quality of Life; Wellbeing; Yoga; Meditation; Psychology
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Heart Failure; Digestive System Diseases; Liver Cirrhosis; Neoplasms; Renal Insufficiency, Chronic; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Waitlist Control (No Intervention)
- Online Program (Experimental): Online program (mindful movement, meditation, breathwork, psychology-based coping skills program)
  Interventions: Behavioral: Online mind-body wellness program
- Online Program + Weekly Check-ins (Experimental): Online program (mindful movement, meditation, breathwork, psychology-based coping skills program) + brief 1-to-1 weekly check-ins with a study team member
  Interventions: Behavioral: Online mind-body wellness program + Weekly Check-ins

INTERVENTIONS:
Behavioral: Online mind-body wellness program — Online program (mindful movement, meditation, breathwork, psychology-based coping skills program)
  Arms: Online Program
Behavioral: Online mind-body wellness program + Weekly Check-ins — Online program (mindful movement, meditation, breathwork, psychology-based coping skills program) + brief weekly check-ins
  Arms: Online Program + Weekly Check-ins

SUMMARY:
Chronic physical conditions are deﬁned as conditions that require ongoing management and treatment over extended periods of time. Chronic physical conditions are not only leading causes of death and disability in North America but they are commonly associated with mental distress and reduced quality of life. Online mind-body wellness programming ranging from physical activity to mindfulness interventions has been shown to be effective in improving mental wellness in a variety of chronic disease populations, but there is a need to evaluate scalable ways to deliver these programs. Building upon a previously developed online wellness program for inﬂammatory bowel disease (IBD) and primary biliary cholangitis (PBC), the research team has developed a mind-body wellness program for adults ≥18 years of age living with different chronic conditions (e.g., cirrhosis, PBC, heart failure). The 12-week program will be delivered online, and include follow- along mindful movement, breathwork and meditation routines, and a psychology based coping skills program. In a three-armed randomized controlled trial, the study will assess the impact on the primary outcome of anxiety and depression as measured through the hospital anxiety and depression scale (HADS). At the beginning and the end of the 12-week research study, participants will complete surveys to assess secondary/exploratory outcome measures including quality of life, fatigue, frailty, demoralization, and healthcare usage.

After the program, the research team will conduct interviews with participants to allow them to share their other feedback about the program. The researchers will also send surveys to the participants eight weeks after the program ends to assess longer- term impacts on primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Identified diagnosis of one of nine chronic conditions (Heart Failure, PBC, Digestive Disease, Cirrhosis, Cancer survivor, Post-transplant, Women who have experienced a cardiac event, Chronic Kidney Disease), or another general category for physical chronic conditions not captured by these nine
* English language proficiency to complete questionnaires and read the educational material
* Access to the Internet and a computer or smart device at home

Exclusion Criteria:

* Receiving compassionate care
* Inability to provide informed written consent
* Severe psychiatric disorders (presence of uncontrolled schizophrenia, post-traumatic stress disorder (PTSD), and/or bipolar disorder unless approved to participate by their physician/psychologist; suicidality nearly every day)
* No access to the internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 825 (Actual)
Dates: Start 2023-02-12 (Actual); Primary Completion 2024-09-22 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 12 weeks
  Depression and anxiety will be measured on the Hospital Anxiety and Depression Scale. The minimum value is 0, the maximum is 21, and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Modified Fatigue Impact Scale (MFIS) | 12 weeks
  The Modified Fatigue Impact Scale (MFIS) assesses the effect of fatigue on cognitive functioning, physical functioning, and psychosocial functioning. The minimum value is 0, the maximum value is 84, and higher scores mean a worse outcome.
Health Related Quality of Life | 12 weeks
  Health related quality of life captured by the quality-of-life Short Form Survey 12 (SF-12). The minimum value is 0, the maximum value is 100, and a higher score means a better outcome.
EQ-5D-5L | 12 weeks
  Cost utility analysis will be facilitated by the EQ-5D-5L which consists of 5- dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) where patients are asked to indicate their health state. The minimum value is 5, the maximum value is 25, and a higher score means a worse outcome.
Capability, Opportunity, Motivation, Behaviour (COM-B) Survey | 12 weeks
  Capability, opportunity, and motivation for behaviour change will be measured on the COM-B survey. The lowest score is 0, the highest score is 60, and higher scores indicate better outcomes.
Satisfaction and Adherence | 12 weeks
  Satisfaction and adherence will be measured using a self-report tool where participants indicate their satisfaction with program elements, and perceived adherence to the program over the study period. The minimum value is 4, the maximum value is 40, and a higher score means a better outcome.

OTHER OUTCOMES:
Demoralization (Exploratory) | 12 weeks
  Demoralization will be captured through self report using the Demoralization Scale-II. The minimum score is 0, the maximum score is 32, and a higher score means a worse outcome.
Edmonton Frail Scale (Exploratory) | 12 weeks
  Frailty will be captured using the Edmonton Frail Scale. The minimum score is 0, the maximum score is 17, and a higher score means a worse outcome.
Fried Frailty (Exploratory) | 12 weeks
  Frailty will be captured using the Fried Frailty Score. The minimum score is 0, the maximum score is 5, and a higher score means a worse outcome.
Healthcare Usage (Exploratory) | 12 weeks
  Healthcare usage will be measured using a self-report tool where participants indicate healthcare service usage during the study period.
Sleep (Exploratory) | 12 weeks
  Impacts on sleep will be captured through self-report using the Patient Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short Form 8a. The minimum score is 8, the maximum score is 56, and a lower score means a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391